CLINICAL TRIAL: NCT02694770
Title: A Phase II Study of Neihulizumab vs "Conventional Treatment" to Treat Steroid-refractory Acute Graft-vs-host Disease (Sr-aGvHD) in Patients Undergoing Allogeneic Hematopoietic Cell Transplantation
Brief Title: A Study Evaluating the Efficacy and Safety of Neihulizumab vs "Conventional Treatment" to Treat Sr-aGvHD
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: corporate decision
Sponsor: AbGenomics B.V Taiwan Branch (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015.011.01
Record Dates: First submitted 2016-02-18; First posted 2016-03-01 (Estimated); Last update posted 2016-04-25 (Estimated); Status verified 2016-04

CONDITIONS: Steroid-refractory aGvHD Subsequent to Allogeneic Hematopoietic Cell Transplantation
Keywords: aGvHD; GvHD; sr-aGvHD; biologics; monoclonal antibody

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Neihulizumab (Experimental): Patients will receive a total of 4 doses of Neihulizumab (AbGn-168H) on Day 1 (Week 0), Day 8 (Week 1), Day 15 (Week 2), and Day 22 (Week 3) by 1-hour i.v. infusion.
  Interventions: Biological: Neihulizumab Treatment
- "Conventional Treatment" (Active Comparator): Patients will receive a 2nd line therapy for aGvHD at the discretion of attending physician according to the standard practice at the study center. Currently there is no treatment for sr-aGvHD is approved in USA or Europe. There is no Standard treatment of this disease is recommended by American Society for Blood and Marrow Transplantation (ASBMT). Therefore, the study is designed to allow any established institutional practice for off-label use of a commercially available product for patients in the Conventional Treatment arm. Patients in this arm may receive treatments provided in ASBMT guidance such as ATG, TNF-alpha inhibitors (such as Etanercept and infliximab), pentostatin, sirolimus, mycophenolate mofetil and extracorporeal photopheresis, methotrexate, basiliximab, daclizumab, inolimomab, denileukin diftitox, alemtuzumab, ATG+ etanercept, Dacliz + etanercept, Dacliz+ infliximab, and Dacliz/inflix/horse ATG.
  Interventions: Biological: Conventional Treatment

INTERVENTIONS:
Biological: Neihulizumab Treatment — Monoclonal antibody
  Other Names: AbGn-168H
  Arms: Neihulizumab
Biological: Conventional Treatment — 2nd line therapy for aGvHD at the discretion of attending physician, including but not limited to biologics such as ATG, TNF-alpha inhibitors, pentostatin, sirolimus, mycophenolate mofetil and extracorporeal photopheresis.
  Arms: "Conventional Treatment"

SUMMARY:
This study is to assess the efficacy of Neihulizumab versus "conventional therapy" and to evaluate safety, pharmacokinetics and immunogenicity in treating steroid-refractory acute Graft-vs-Host Disease

DETAILED DESCRIPTION:
This current Phase II trial is a randomized, open label, controlled, multiple dose, multi-centre study to study the clinical efficacy and safety of Neihulizumab vs "Conventional Treatment" to treat steroid-refractory acute graft-vs-host disease (sr-aGvHD) in patients undergoing allogeneic hematopoietic cell transplantation.

This study will enroll a minimum of 90 patients, approximately 60 in Neihulizumab treatment arm and 30 in Conventional treatment control arm.

The primary objectives is to evaluate the efficacy of Neihulizumab treatment in patients with steroid-refractory acute GvHD compared to "conventional treatment." The secondary objectives are to investigate safety, pharmacokinetics, and immunogenicity of Neihulizumab administration in subjects with steroid-refractory acute GvHD.

For safety evaluation, the parameters to be assessed are adverse events (AEs), discontinuation of therapy due to AEs, safety laboratory analysis, ECG, vital signs, physical examination, and immunogenicity.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must be ≥18years of age, males or females;
2. Patient must have been recipients of a single allogeneic HCT; bone marrow, peripheral blood and/or umbilical cord blood recipients are allowed
3. Patients must have aGvHD without feature of classic chronic GvHD or overlap GvHD;
4. Patients must have received no prior treatment for aGvHD other than steroids;
5. Patients must have biopsy proven grade II to IV aGvHD progressing after at least 3 days, non-improving grade III to IV aGvHD persistent after at least 7 days, or non-improving grade II aGvHD persistent after at least 14 days of methylprednisolone 2mg/kg/day or equivalent; Patients with initial response but have flare of aGvHD within 14 days with methylprednisolone > 0.5 mg/kg/day or equivalent are also eligible;
6. Patient must have an ANC of > 500/mm3 and no evidence of HCT graft failure or multi-organ failure;
7. Patient must have Karnofsky Performance Status (KPS) ≥50%;
8. Patient must give informed consent and sign an approved consent form prior to any study procedures;
9. Females of childbearing potential must have a negative pregnancy test result prior to enrollment. Males and females of childbearing potential must agree to use a highly effective method of birth control during the study.

Exclusion Criteria:

1. Uncontrolled infections not responsive to antimicrobial therapy or requiring intensive critical care or vasopressors;
2. Evidence of end-organ infection due to CMV;
3. HIV infection or a known HIV-related malignancy (NOTE: patients positive for hepatitis B or hepatitis C are not excluded, and may be evaluated on a case by case basis).
4. Tuberculosis, history of tuberculosis or a known positive Quantiferon test for tuberculosis
5. Donor lymphocyte infusion for residual or relapsed disease or mixed chimerism. DLI as part of the planned HCT protocol are allowed
6. Relapsed disease after transplant or progressive malignant disease, including post-transplant lymphoproliferative disease; any secondary malignancy diagnosed since HCT
7. Renal failure requiring hemodialysis
8. Need ICU care, with life expectancy of less than 28 days, with ongoing or unresolved veno-occlusive disease, with unstable hemodynamics, with evidence of current or previous clinically significant disease, medical condition or finding of the medical examination (including vital signs and ECG), that in the opinion of the Investigator, would compromise the safety of the patient or the quality of the data
9. History of allergy/hypersensitivity to a systemically administered biologic agent or its excipients
10. Pregnant or nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-07; Primary Completion 2017-09 (Estimated); Study Completion 2018-02 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (Complete Response+Partial Response) | Day 28 after the initiation of sr-aGvHD treatment

SECONDARY OUTCOMES:
Overall response rate (Complete Response+Partial Response) | Day 56 after the initiation of sr-aGvHD treatment
Complete Response+Very Good Partial Response | Day 28 and Day 56 after the initiation of sr-aGvHD treatment
Overall survival | Day 180 after the initiation of sr-aGvHD treatment
Cumulative steroid dose | Day 28 after the initiation of sr-aGvHD treatment
Cumulative incidence of chronic GvHD | Day 180 after the initiation of sr-aGvHD treatment
Cumulative incidence of primary disease relapse | Day 180 after the initiation of sr-aGvHD treatment

CONTACTS AND LOCATIONS:
Overall Officials: Shih-Yao Lin, MD, PhD, Study Chair — AbGenomics B.V.; Paul Martin (Lead), MD, Principal Investigator — Fred Hutchinson Cancer Center; Marco Mielcarek (Co-Lead), MD, Principal Investigator — Fred Hutchinson Cancer Center; Amin Alousi (Co-Lead), MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (2):
- United States (2):
  - MD Anderson Cancer Center, Houston, Texas
  - Fred Hutchinson Cancer Research Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No